CLINICAL TRIAL: NCT01074866
Title: The Effects of Neurally Adjusted Ventilatory Assist (NAVA) on Improving Patient-ventilator Interaction in Patients Undergoing Ventilation for Acute Respiratory Failure
Brief Title: Neurally Adjusted Ventilatory Assist for Non Invasive Ventilation and Patient-ventilator Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University Hospital St Luc, Brussels (Other); University Hospital Sart Tilman, Liege (Unknown); University of Lausanne Hospitals (Other); Notre Dame de Grace Hospital, Gosselies (Unknown)
Responsible Party: Intensive Care Unit, HUG, University hospital of Geneva
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: NAVA_NIV
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2010-01

CONDITIONS: Non Invasive Ventilation; Patient Ventilator Interaction
Keywords: Mechanical ventilation; Non invasive Ventilation; Patient-ventilator interaction; Pressure support; Neurally adjusted ventilatory assist
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure support (No Intervention): Non invasive ventilation under pressure support (PS)
- Neurally Adjusted Ventilatory Assist (Active Comparator): Non invasive ventilation under Neurally Adjusted ventilatory Assist
  Interventions: Device: Neurally Adjusted Ventilatory Assist

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist — Non invasive ventilation under Neurally adjusted Ventilatory Assist
  Other Names: NAVA
  Arms: Neurally Adjusted Ventilatory Assist

SUMMARY:
The present study aims to compare various parameters reflecting patient-ventilator synchrony during standard pressure support (PS) and Neurally Adjusted Ventilatory assist (NAVA) in a group of patients receiving non invasive ventilation (NIV)for an episode of acute respiratory failure of various origin.

DETAILED DESCRIPTION:
The present study aims to compare various parameters reflecting patient-ventilator synchrony during standard pressure support (PS) and Neurally Adjusted Ventilatory assist (NAVA) in a group of patients receiving non invasive ventilation (NIV)for an episode of acute respiratory failure of various origin. The subgroup of COPD patients will be analyzed separately. The effects of various setting of Neurally adjusted ventilatory assist on patient-ventilator interaction will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU and treated with Non invasive ventilation for acute respiratory failure of any origin

Exclusion Criteria:

* severe hypoxemia requiring an FIO2>0.6
* hemodynamic instability
* known oesophageal problem
* active upper gastro-intestinal bleeding
* any other contraindication to the insertion of a naso-gastric tube
* impaired consciousness or absence of patient cooperation
* facial or laryngeal lesions contraindicating the use of NIV
* poor short term prognosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Patient-ventilator synchronization parameters

CONTACTS AND LOCATIONS:
Overall Officials: Didier Tassaux, MD, Study Director — HUG, University hospital Geneva
Locations (4):
- Belgium (2):
  - St Luc University hospital, Brussels
  - Bernard Lambermont, Liège
- Switzerland (2):
  - HUG, University Hospital, Geneva
  - CHUV University hospital of Lausanne, Lausanne